CLINICAL TRIAL: NCT04182698
Title: Phase I / II Clinical Study on the Safety and Preliminary Efficacy of Anlotinib Hydrochloride Combined With Platinum-containing Simultaneous Radiotherapy in the Treatment of Locally Advanced Non-small Cell Lung Cancer
Brief Title: Study of Anlotinib Plus Chemoradiotherapy in Patients With Locally Advanced NSCLC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Collaborators: Tang-Du Hospital (Other); Xijing Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Shaanxi Provincial Cancer Hospital (Other); Shaanxi Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SecondXianJiaotongU2
Record Dates: First submitted 2019-11-22; First posted 2019-12-02 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Patients With Non-small Cell Lung Cancer
Keywords: Alotinib non-small cell lung cancer

STUDY DESIGN:
Intervention Model Description: Experimental group: anlotinib (D1-14, d22-36, followed by 21 days cycle, taking medicine for 2 weeks, stopping for 1 week).
  Group 1: 8mg po qd, Group 2: 10mg po qd, Group 3: 12mg po qd;
  Combined chemotherapy:
  Cisplatin + etoposide or PC: carboplatin AUC2, paclitaxel 45-50 mg 2 per week; Cisplatin + pemetrexed (non-squamous cell carcinoma). Simultaneous radiotherapy: 3D-CRT or IMRT external radiotherapy (60-66 Gy, 2.0 Gy / day).
  The curative effect was evaluated after 6 weeks of simultaneous radiotherapy and chemotherapy combined with alotinib, and then the efficacy of alotinib or chemotherapy was maintained until PD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Experimental group: anlotinib(d1-14, d22-36), followed by 21 days period, 2 weeks medication, 1 week maintenance therapy.
  . Group II: 10 mg po qd, Group III: 12 mg po qd;
  Combined chemotherapy:
  Cisplatin + etoposide Or PC: carboplatin AUC2, paclitaxel 45-50 mg 2 per week; Cisplatin + cultured beauty (non squamous cell carcinoma). Synchrotron radiation: radiotherapy combined with radiotherapy (3D-CRT or IMRT) (60-66Gy / day).
  The curative effect was evaluated after 6 weeks of simultaneous radiotherapy and chemotherapy combined with alotinib, and then the efficacy of alotinib or chemotherapy was maintained until PD.
  Interventions: Drug: Simultaneous chemoradiotherapy for An Luo

INTERVENTIONS:
Drug: Simultaneous chemoradiotherapy for An Luo — Experimental group: anlotinib(d1-14, d22-36), followed by 21 days period, 2 weeks medication, 1 week maintenance therapy.
  . Group II: 10 mg po qd, Group III: 12 mg po qd;
  Combined chemotherapy:
  Cisplatin + etoposide Or PC: carboplatin AUC2, paclitaxel 45-50 mg 2 per week; Cisplatin + cultured beauty (non squamous cell carcinoma). Synchrotron radiation: radiotherapy combined with radiotherapy (3D-CRT or IMRT) (60-66Gy / day).
  The curative effect was evaluated after 6 weeks of simultaneous radiotherapy and chemotherapy combined with alotinib, and then the efficacy of alotinib or chemotherapy was maintained until PD.

SUMMARY:
Lung cancer is the most common cancer, accounting for 20% of cancer-related deaths worldwide. In 2015, an estimated 610,200 patients (22 per cent of cancer-related deaths) died of lung cancer. Non-small cell lung cancer ((NSCLC)) accounts for 80% to 85% of lung cancer. Most patients are locally advanced or metastatic diseases at the time of diagnosis. Some IIIA tumors are considered resectable, but many IIIA (with larger N2) and IIIB (T4, any NM0, any TN3M0) are not considered suitable for surgery. Since the 1990s, simultaneous radiotherapy and chemotherapy ((CHRT)) has become the cornerstone of (NSCLC) in locally advanced non-small cell lung cancer (NSCLC). At present, there is no clinical evidence of survival benefits of synchronous radiotherapy plus TKI targeted therapy for unresectable stage Ⅲ A and stage Ⅲ B non-small cell lung cancer. However, a HELPER STUDY study was conducted to evaluate the efficacy and safety of continuous intravenous infusion combined with EP regimen plus concurrent radiotherapy in the treatment of unresectable stage Ⅲ NSCLC. The median survival time was 34.7 months and the 3-year survival rate was 47.7%. Anlotinib capsule is a small molecule multi-target tyrosine kinase inhibitor. This is a single group partitioned, multicenter, exploratory clinical study to observe and evaluate the safety and tolerance of anlotinib hydrochloride combined with cisplatin plus etoposide or pemetrexed in the treatment of locally advanced NSCLC patients. To determine the maximum tolerable dose of (MTD) and / or stage II clinical recommended dose (RP2D) and evaluate its preliminary efficacy. In the first stage of this study, 12 patients with locally advanced NSCLC were divided into 3 experimental groups. After taking three different doses of anlotinib combined with platinum simultaneous radiotherapy, the dose limited toxicity was observed, and the maximum tolerable dose was determined in the second stage. 78 patients were enrolled according to RP2D, and the indexes such as ORR were evaluated. To evaluate the safety and efficacy of anlotinib combined with platinum-containing simultaneous radiotherapy in the treatment of locally advanced NSCLC.

Anlotinib (D1-14, d22-36, followed by a 21-day cycle, taking medicine for 2 weeks, stopping for 1 week).

Group 1: 8mg po qd, Group 2: 10mg po qd, Group 3: 12mg po qd;

Combined chemotherapy:

Cisplatin + etoposide Or PC: carboplatin AUC2, paclitaxel 45-50 mg 2 per week; Cisplatin + pemetrexed (non-squamous cell carcinoma). Simultaneous radiotherapy: 3D-CRT or IMRT external radiotherapy (60-66 Gy, 2.0 Gy / day).

The curative effect was evaluated after 6 weeks of simultaneous radiotherapy and chemotherapy combined with alotinib, and then the efficacy of alotinib or chemotherapy was maintained until PD.

Main outcome measures:

Phase I main outcome measures: maximum tolerated dose (MTD), dose limited toxic (DLT).

Main indicators of II: objective remission rate (ORR). Secondary indicators: disease control rate (DCR), progression-free survival (PFS)

DETAILED DESCRIPTION:
Lung cancer is the most common cancer, accounting for 20% of cancer-related deaths worldwide. In 2015, an estimated 610,200 patients (22 per cent of cancer-related deaths) died of lung cancer. Non-small cell lung cancer ((NSCLC)) accounts for 80% to 85% of lung cancer. Most patients are locally advanced or metastatic diseases at the time of diagnosis. Some IIIA tumors are considered resectable, but many IIIA (with larger N2) and IIIB (T4, any NM0, any TN3M0) are not considered suitable for surgery.

Since the 1990s, simultaneous radiotherapy and chemotherapy ((CHRT)) has become the cornerstone of (NSCLC) in locally advanced non-small cell lung cancer (NSCLC). At present, there is no clinical evidence of survival benefits of synchronous radiotherapy plus TKI targeted therapy for unresectable stage Ⅲ A and stage Ⅲ B non-small cell lung cancer. However, a HELPER STUDY study was conducted to evaluate the efficacy and safety of continuous intravenous infusion combined with EP regimen plus concurrent radiotherapy in the treatment of unresectable stage Ⅲ NSCLC. The median survival time was 34.7 months and the 3-year survival rate was 47.7%. anlotinib capsule is a small molecule multi-target tyrosine kinase inhibitor. Compared with bevacizumab, its anti-tumor therapy has three unique advantages: 1. Inhibition of multiple targets, such as VEGFR, PDGFR, FGFR, c-Kit, etc., improves the effectiveness against a variety of malignant tumors, mainly in the following three aspects: first, it is aimed at several fatal pathways of tumor cells themselves, namely, driving gene pathways. Seal them all off one by one; Secondly, blocking vascular targeting: inhibition of vascular endothelial cell receptors such as VEGFR, PDGFR, FGFR and so on. These three tyrosine kinase receptors and their corresponding ligands play an important role in angiogenesis: VEGF can proliferate cells, FGF and PDGF make vascular endothelial cells chemotactic to the vicinity of the tumor to form neovascularization. Let the pericytes of the blood vessels be covered to form a complete structure of the blood vessels; Finally, it can inhibit both tumor cells and tumor angiogenesis: because only suppressing tumor growth, tumor cells secrete some factors to save themselves, resulting in dense compensation for the vascular network, so that the tumor is supplied with blood. Will madly proliferate again, forming drug-resistant tumors. two。. Oral drug, convenient and effective: pharmacokinetic studies on the metabolism of anlotinib in vivo have found that the peak time of the drug in blood is 4 to 11 hours after administration, and the half-life is about 90 hours. Stopping for one week for two weeks can keep the blood drug concentration in the treatment window stably, which is safe and effective, more tolerant, convenient to use, and can improve the quality of life of patients. 3. Compared with the macromolecular monoclonal antibody represented by bevacizumab, the half-life of the drug is shorter, the long-term use of TKI, is smaller, the corresponding side effects are less, and the incidence of adverse events is lower than that of bevacizumab. In the II phase study of erlotinib combined with bevazumab, the incidence of hypertension with JO25567,3 degree or above was as high as 60%, and the tolerance of the patients was relatively poor. In the ALTER 0303 test, the common adverse reactions in the anlotinib group were fatigue, hypertension, skin toxicity and so on, but the incidence of grade 1-2 AE,SAE was lower (15.3%). And most of them can be relieved by symptomatic treatment or reduction, and the safety of the drug is good. This study was a clinical study on the treatment of locally advanced unresectable NSCLC with anlotinib hydrochloride combined with platinum-containing simultaneous radiotherapy. To observe and evaluate the safety and tolerance of anlotinib hydrochloride combined with cisplatin plus etoposide or pemetrexed in the treatment of locally advanced NSCLC patients. To determine the maximum tolerable dose of (MTD) and / or stage II clinical recommended dose (RP2D) and evaluate its preliminary efficacy. In the first stage of this study, 12 patients with locally advanced NSCLC were divided into 3 experimental groups. After taking three different doses of anlotinib combined with platinum simultaneous radiotherapy, the dose limited toxicity was observed, and the maximum tolerable dose was determined in the second stage. 78 patients were enrolled according to RP2D, and the indexes such as ORR were evaluated. To evaluate the safety and efficacy of anlotinib combined with platinum-containing simultaneous radiotherapy in the treatment of locally advanced NSCLC.

1. Administration regimen: anlotinib (21 days as a cycle, 2 weeks, 1 week). Group 1: 8mg po qd, Group 2: 10mg po qd, Group 3: 12mg po qd;

   Combined chemotherapy:

   Cisplatin 50 mg 2, ivgt, D1, 8, 29, 36, etoposide 50 mg 2, ivgt, D1-5, 29-33; Or PC: carboplatin AUC2, paclitaxel 45-50 mg 2 per week; Cisplatin 25 mg 2, ivgt, D1-3, 22-24, pemetrexed ivgtt,500 mg/m2,ivgtt,d1, d22; (non-squamous cell carcinoma).

   Simultaneous radiotherapy: 3D-CRT or IMRT external radiotherapy (60-66 Gy, 2.0 Gy / day).

   The curative effect was evaluated after 6 weeks of simultaneous radiotherapy and chemotherapy combined with alotinib, and then the efficacy of alotinib or chemotherapy was maintained until PD.
2. Observation index.

   Main outcome measures:

   Phase I main outcome measures: maximum tolerated dose (MTD), dose limited toxic (DLT).

   Main indicators of II: objective remission rate (ORR). Secondary indicators: disease control rate (DCR), progression-free survival (PFS).
3. Administration cycle: patients with complete remission of (CR), partial remission of (PR) and stable (SD) continued to give drugs until disease progression (PD), intolerable toxicity or patients asked for withdrawal or progression of (PD).
4. Effectiveness evaluation and analysis: effectiveness evaluation is conducted every two cycles (the time is based on the number of calendar days and is not affected by drug withdrawal), and the evaluation time is within 7 days of the end of the cycle (except statutory holidays). CT should be performed in the evaluation (CT evaluation is recommended every two cycles and PET-CT evaluation is performed once a year). The imaging techniques used in the evaluation of the same patient should be the same, and all imaging data should be retained.5. Treatment of possible toxic and side effects of anlotinib hydrochloride.

The results of phase I anlotinib monotherapy tolerance test showed that the main adverse reactions associated with alrotinib hydrochloride were hand and foot syndrome, hypertension, albuminuria, diarrhea, gastrointestinal bleeding, thrombocytopenia and albuminuria, hyperlipidemia. Hyperglycemia and so on.

5.1 hand and foot Syndrome (Palmar-plantar erythrodysesthesia syndrome)). Hand and foot syndrome is palm-foot sensation dull or limb turn red, obvious discomfort, swelling, tingling, pressure or stress area performance is more obvious. Tumor patients can occur during chemotherapy or molecular targeted therapy. Grade 1 showed painless mild skin changes or dermatitis (such as erythema, edema, hyperkeratosis), grade 2 showed painful skin changes (such as exfoliation, blisters, bleeding, swelling, excessive keratosis). Affect tool daily life activities; Grade 3 showed severe skin changes (exfoliation, blistering, bleeding, edema, hyperkeratosis) with pain and affected personal activities of daily life.

For patients with grade 1 toxicity, there is often no need for support treatment, grade 2 or above toxic patients consider the following symptomatic support treatment: including: strengthen skin care, keep the skin clean, avoid secondary infection, avoid pressure or friction; Use moisturizing creams or lubricants, topical lotions or lubricants containing urea and corticosteroids, and local antifungal or antibiotic treatments if necessary.

5.2 Hypertension. Blood pressure should be monitored daily for the first 6 weeks of this study. If there is an increase in blood pressure, it is necessary to actively communicate with the doctor. When blood pressure rises, conventional antihypertensive therapy can be controlled. For uncontrollable increases in blood pressure, they can also be alleviated by reducing the amount of targeted drugs or stopping them.

Suggestions on staging and routine treatment of hypertension.

Hypertension refers to a pathological increase in blood pressure, which is repeatedly measured over and over 140/90mmHg. Severity rating:

Grade 1: prehypertension (systolic blood pressure 120-139, diastolic blood pressure 80-89 mmHg) there is no indication of antihypertensive drugs, only blood pressure is monitored. Grade 2: the first stage of hypertension (systolic blood pressure 140159mmHg, diastolic blood pressure 90-99mmHg), the need for medical intervention, repeated or lasting (greater than or equal to 24 hours), symptomatic systolic blood pressure increased more than 20mmHg or the previous normal range increased more than 140mmHg; Blood pressure needs to be monitored with single drug treatment, and most of them use thiazide diuretics, but also consider angiotensin converting enzyme inhibitor (ACEI), angiotensin Ⅱ receptor blocker (ARB), β receptor blocker and calcium channel blocker. Stage 3: stage II hypertension (systolic blood pressure greater than or equal to 160mm Hg and diastolic blood pressure greater than or equal to 100mmHg); requires medical intervention; requires a variety of drugs, usually thiazide diuretics and ACEI or beta blockers or calcium channel blockers. Level 4: life-threatening (e.g. malignant hypertension, transient or persistent nerve damage, hypertension crisis); requires emergency treatment. At present, there is no unified classification at home and abroad. Recently, it has been divided into two types from the point of view of clinical treatment.

The main results are as follows: (1) hypertensive emergency (Hypertension emergencies), diastolic pressure > 120 mmHg, is associated with acute or progressive target organ damage, such as cerebral infarction, intracranial or subarachnoid hemorrhage, hypertensive encephalopathy, etc. Among them, progressive or rapid hypertension based on chronic essential hypertension was the most common (about 40% to 50%).

(2) (Hypertension urgencies), diastolic blood pressure > 120 mmHg in hypertensive emergency was not accompanied by or only slight organ damage.

Sodium nitroprusside or nifedipine was used to reduce blood pressure rapidly, diazepam and phenobarbital were used to stop convulsions, furosemide and mannitol were dehydrated, sodium excretion and intracranial pressure were reduced.

In the event of hypertension crisis, the patient should stop taking the drug and withdraw from this clinical study.

5.3 treatment of diarrhoea. Patients with grade 1 or 2 diarrhea can be given supportive treatment, such as the earliest onset of Lopebutylamine (such as oral administration of 4 mg, and then oral 2mg every 2 hours until diarrhea is relieved).

5.4 Management of Digestive tract Hemorrhage. Gastrointestinal bleeding, including fecal occult blood (+ +), hematemesis or bloody stool, should be treated actively. Patients with upper gastrointestinal bleeding should fast, stop acid, protect gastric mucosa, stop bleeding (hemostatic cyclic acid, standing hemostasis, etc.), transfusion and supporting treatment, and octreotide can be used if necessary. Patients with lower gastrointestinal bleeding should be given hemostasis, blood transfusion and supporting treatment, etc.; if the bleeding is uncontrollable, surgical assistance should be requested.

5.5 suggestions for the treatment of albuminuria. During the whole period of treatment, proteinuria was closely monitored in all patients, and 24-hour urinary protein determination should be performed in those with a history of hypertension and two consecutive times of urinary protein ≥ + +.

After the occurrence of albuminuria, the principles of dose adjustment are as follows: urinary protein + or < 3g/24h continue to be given according to the plan and symptomatic treatment; If albuminuria ≥ 3G for 24 hours, the administration was suspended and treated symptomatically until the urine protein < 3g/24h lowered a dose level and continued to be administered. If the dose is reduced, the second occurrence of urinary protein ≥ 3g 24 hours, can be restored to < 3g/24h and then reduced by one dose level of treatment. However, if the third occurrence of urinary protein ≥ 3g 24h, the test would be terminated.

If 4 degrees proteinuria (nephrotic syndrome) occurs, the drug will be permanently discontinued and withdrawn from this clinical study.

5.6 Management of hyperlipidemia and hyperglycemia. The pre-treatment state and eating habits of patients with hyperlipidemia should be taken into account. In addition to diet, grade 2 or higher hypercholesterolemia (≥ 7.75mmol/L), or grade 2 or higher hypertriglyceridemia (≥ 2.5 times the normal upper limit), HMG-CoA reductase inhibitors (atorvastatin, etc.) or appropriate lipid-lowering drugs should be used.

Dose adjustment of anlotinib hydrochloride. In the event of drug-related toxicity, the toxicity was graded according to NCI CTCAE (version 4.0).

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 70 years old; two。. Histologically or cytologically confirmed, locally advanced IIIA 、IIIB or IIIC NSCLC (according to version 8); 3.ECOG score: 0-1; 4. Those who have not received targeted and immunotherapy in the past; 5. Patients who had not undergone surgery in the past; 6. The damage caused by other treatments was recovered, in which the interval of receiving nitroso or mitomycin was ≥ 6 weeks, receiving other cytotoxic drugs and bevacizumab (Avastin) ≥ 4 weeks; 7. The function of the main organs is normal, that is, the following criteria are met:

1. the standard of blood routine examination should be met (no blood transfusion and blood products within 14 days, not corrected by G-CSF and other hematopoietic stimulating factors): A. HB ≥ 90g; B. ANC ≥ 1.5 × 109; C. PLT ≥ 80 × 109;
2. biochemical tests shall meet the following criteria: A. TBIL < 1.5ULN; B. ALT and AST < 2.5ULN; c. Serum Cr ≤ 1.5ULN or endogenous creatinine clearance > 50 ml/min (Cockcroft-Gault formula); 8. Doppler Echocardiography: left Ventricular ejection fraction (LVEF) ≥ 50% normal Lower limit (LLN).

9. The subjects volunteered to join the study and signed an informed consent form with good compliance and follow-up.

Exclusion Criteria:

1. Small cell lung cancer (including small cell carcinoma and non-small cell carcinoma mixed lung cancer); The patients with positive mutations of 2.EGFR, ALK and ROS1 genes were feasible for targeted therapy.

3. In the past, more than 4 cycles of chemotherapy were received. 4. Hemoptysis in patients with non-small cell lung cancer (> 50 mL / day), tumor with cavity or necrosis; 5. The imaging showed that the important blood vessels had been invaded by the tumor or the researchers determined that the tumor might invade the important blood vessels during the follow-up period and cause fatal bleeding.

6. Those with hypertension and could not be reduced to the normal range after antihypertensive drug treatment (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg);) had a history of unstable angina pectoris. Patients with newly diagnosed angina pectoris within 3 months before screening or myocardial infarction events within 6 months before screening, arrhythmias (including QTcF ≥ 470 ms) required long-term use of antiarrhythmic drugs and New York Heart Association grade ≥ II cardiac insufficiency.

7. It has obvious factors affecting oral drug absorption, such as inability to swallow, chronic diarrhea and intestinal obstruction.

8. Patients with abnormal coagulation function (INR > 1.5 or prothrombin time (PT) > ULN+ 4 seconds or APTT > 1.5 ULN),) had bleeding tendency or were treated with anticoagulants or vitamin K antagonists such as warfarin, heparin or their analogues. On the premise that the international standardized ratio of prothrombin time (INR) ≤ 1.5, low dose heparin (6000U / d for adults) or low dose aspirin (not exceeding 100U / d) is allowed.

9. Urine routine showed that urinary protein ≥ + +, or 24-hour urinary protein quantity ≥ 1.0g; 10. The bleeding symptoms in the first 3 months have obvious clinical significance or definite bleeding tendency, such as gastrointestinal bleeding, hemorrhagic ulcer, positive fecal occult blood, etc.

11. There were venous thromboembolism events in the first 12 months, such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep venous thrombosis and pulmonary embolism.

twelve。. The patients participated in clinical trials of other antineoplastic drugs within 4 weeks.

The researchers judged other situations that may affect the conduct of clinical studies and the determination of the results of the studies.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-11-22 (Estimated); Primary Completion 2021-05-17 (Estimated); Study Completion 2021-05-17 (Estimated)

PRIMARY OUTCOMES:
ORR (Objective control rate) | approximately 18 months
  complete response(CR)+partial response(PR) according to RECIST 1.1

SECONDARY OUTCOMES:
OS (Overall survival) | approximately over 3-5 years
  overall survival is defined as the time from randomization to death from any cause
PFS (Progression-Free survival) | approximately 36 months
  progression-free survival is defined as the time from enrollment to the date of first document disease progression or death from any cause
DCR (Disease control rate) | approximately 18 months
  The rate of CR, PR plus SD

CONTACTS AND LOCATIONS:
Locations (1):
- The second affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller KD, Siegel RL, Lin CC, Mariotto AB, Kramer JL, Rowland JH, Stein KD, Alteri R, Jemal A. Cancer treatment and survivorship statistics, 2016. CA Cancer J Clin. 2016 Jul;66(4):271-89. doi: 10.3322/caac.21349. Epub 2016 Jun 2. PMID 27253694
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Liang J, Bi N, Wu S, Chen M, Lv C, Zhao L, Shi A, Jiang W, Xu Y, Zhou Z, Wang W, Chen D, Hui Z, Lv J, Zhang H, Feng Q, Xiao Z, Wang X, Liu L, Zhang T, Du L, Chen W, Shyr Y, Yin W, Li J, He J, Wang L. Etoposide and cisplatin versus paclitaxel and carboplatin with concurrent thoracic radiotherapy in unresectable stage III non-small cell lung cancer: a multicenter randomized phase III trial. Ann Oncol. 2017 Apr 1;28(4):777-783. doi: 10.1093/annonc/mdx009. PMID 28137739
- [Background] Han B, Li K, Wang Q, Zhang L, Shi J, Wang Z, Cheng Y, He J, Shi Y, Zhao Y, Yu H, Zhao Y, Chen W, Luo Y, Wu L, Wang X, Pirker R, Nan K, Jin F, Dong J, Li B, Sun Y. Effect of Anlotinib as a Third-Line or Further Treatment on Overall Survival of Patients With Advanced Non-Small Cell Lung Cancer: The ALTER 0303 Phase 3 Randomized Clinical Trial. JAMA Oncol. 2018 Nov 1;4(11):1569-1575. doi: 10.1001/jamaoncol.2018.3039. PMID 30098152
- [Background] Lin Y, Zhai E, Liao B, Xu L, Zhang X, Peng S, He Y, Cai S, Zeng Z, Chen M. Autocrine VEGF signaling promotes cell proliferation through a PLC-dependent pathway and modulates Apatinib treatment efficacy in gastric cancer. Oncotarget. 2017 Feb 14;8(7):11990-12002. doi: 10.18632/oncotarget.14467. PMID 28061477
- [Background] Hu M, Hu Y, He J, Li B. Prognostic Value of Basic Fibroblast Growth Factor (bFGF) in Lung Cancer: A Systematic Review with Meta-Analysis. PLoS One. 2016 Jan 29;11(1):e0147374. doi: 10.1371/journal.pone.0147374. eCollection 2016. PMID 26824699
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5355320/
- See also: Related Info — https://journals.plos.org/plosone/article?id=10.1371/journal.pone.0147374